CLINICAL TRIAL: NCT00000108
Title: Effects of Training Intensity on the CHD Risk Factors in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: NCRR-M01RR00042-1647; M01RR000042 (NIH)
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Cardiovascular Diseases; Coronary Disease
Keywords: exercise
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Motor Activity | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
The purpose of this research is to find out whether training at different exercise intensities reduces the risk of developing cardiovascular disease (CVD) to a different extent. Heart attacks and stroke are the leading cause of death in older women. Reduced variability of the heart rate and increased dips and swings in blood pressure are risks factors that predict the chance of developing CVD as are increased levels of clotting protein fibrinogen and plasminogen activator inhibitor 1, and high levels of LDL-cholesterol (>160mg/dl). We will be measuring all of these risk factors and any changes in your body fat level before you start training and after 15 and 30 weeks of training in the form of walking. At the present time the effects of exercise intensity on these factors are not well understood. This study will add to the basic understanding of these issues and allow us to recommend to postmenopausal women optimal exercise intensities to lose body fat and reduce the risk of developing CVD.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal and preferably on hormone replacement therapy
* In good general health
* Have a body mass index (BMI, weight in kg/height in m2) of between 25 and 40
* Exercise less than 20 min/day two days a week

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- 3060G Central Campus Recreation Bldg 401 Washtenaw Ave., Ann Arbor, Michigan, United States